CLINICAL TRIAL: NCT06471114
Title: Evaluation of the Efficacy of Systemic Treatments for Alopecia
Brief Title: Evaluation of the Efficacy of Systemic Treatments for Alopecia (ESTAA)
Acronym: ESTAA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0239 - ESTAA
Record Dates: First submitted 2024-04-29; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-10

CONDITIONS: Alopecia Areata
Keywords: severe
MeSH Terms: conditions — Alopecia Areata; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study was to retrospectively assess the efficacy and safety of systemic treatments in patients with alopecia areata, by recruiting cases from the HUGO network (Hôpitaux Universitaires du Grand Ouest), a network of 5 hospitals : Brest, Nantes, Rennes, Angers and Tours.

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe alopecia
* Has received at least one systemic treatment for at least 3 months (among methotrexate, intravenous or oral corticosteroid therapy, Ciclosporin, UVA/UVB phototherapy)
* Patient affiliated to a social security scheme
* Age greater than or equal to 18 years

Exclusion Criteria:

* Patients under legal protection (guardianship, curatorship, etc.)
* Refusal to participate
* Other cause of alopecia
* Follow-up less than 3 months
* Age under 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients selected from 5 university hospitals in the HUGO network (Brest, Rennes, Tours, Angers, Nantes).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Short-term efficacy and security of systemic treatments | From January 2010 to December 2020
  Response rates including complete response or partial response or no response for each modality of treatment. and Side effects rate

SECONDARY OUTCOMES:
Long-term efficacy of systemic treatments | From January 2010 to December 2020
  Among responders (CR and PR), the maintained response rate and relapse rate

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement